CLINICAL TRIAL: NCT00271544
Title: Attain Model 4196 Left Ventricular (LV) Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: 4196 Clinical Trial Leader, Medtronic, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 241
Record Dates: First submitted 2005-12-28; First posted 2006-01-02 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac pacing; left ventricular lead; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4196 Lead (Experimental): Non-randomized study.
  Interventions: Device: Pacing Lead

INTERVENTIONS:
Device: Pacing Lead — implant and follow-up of study device

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy (CRT) may be prescribed. CRT is similar to a pacemaker. It is placed (implanted) under the skin of the upper chest. CRT is delivered as tiny electrical pulses to the right and left ventricles through three or four leads (flexible insulated wires) that are inserted through the veins to the heart. The purpose of this study is to evaluate a new lead for delivering energy to the left ventricle (bottom left chamber of the heart).

ELIGIBILITY:
Inclusion Criteria:

* QRS greater than or equal to 120 milliseconds (The QRS interval is a measurement of how the electrical signal involved in a heart beat travels, or is conducted, through the ventricles. A wide QRS (more than 120) suggests that there is a conduction problem, or block, in the ventricles.)
* Left Ventricular Ejection Fraction (EF) less than or equal to 35 percent (Ejection Fraction is a measurement of how well the left ventricle pumps blood out to the rest of the body. The higher the EF the more blood the ventricle is pumping.)
* Subject has moderate to severe heart failure despite medications

Exclusion Criteria:

* Subjects with a previous lead in the left ventricle or previous implant attempt within 30 days of implant or ongoing complications from a previous unsuccessful attempt
* Subjects with chest pain or who have had a heart attack within the past month before enrollment in the study
* Subjects that have had certain surgeries on their heart within the past three months
* Subjects with chronic (permanent) fast heart beats in the upper chambers of the heart (atrial arrhythmias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2007-02; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ramza, MD, PHD, Principal Investigator — St. Luke's Mid America Heart Institute, Kansas City MO
Locations (24):
- United States (19):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Long Beach, California
  - Palo Alto, California
  - Davenport, Iowa
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Raleigh, North Carolina
  - Mayfield Heights, Ohio
  - Wynnewood, Pennsylvania
  - Spartanburg, South Carolina
  - Kingsport, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Burlington, Vermont
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of patients enrolled after meeting inclusion/exclusion criteria was 190. Total number of patients that received an implant attempt was 186. Total number of patients with a 4196 lead attempt was 177. Total number of patients successfully implanted with a 4196 lead was 170. Some data was not reported and deviations were recorded.
Groups:
- 4196 Lead: Subjects underwent Model 4196 left ventricular lead implant attempt
Period: Overall Study
Arm/Group | 4196 Lead
Started | 190 (Total number of subjects enrolled.)
Implant Attempted | 186 (Total number of subjects completed baseline and underwent system implant attempt.)
Model 4196 Lead Attempted | 177 (Total number of subjects attempted Model 4196 lead.)
Completed | 170 (Total number subjects successfully implanted 4196 lead.)
Not Completed | 20
Not completed — Subjects did not receive a 4196 lead | 7
Not completed — Model 4196 lead not attempted | 9
Not completed — Implant not attempted | 4

BASELINE CHARACTERISTICS:
Arm/Group | 4196 Lead
Number analyzed (Participants) | 186
Age, Categorical [Count of Participants; unit: Participants] — All subjects who underwent an implant attempt (186) were included in the study population analyses.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 57
    >=65 years | 129
Age Continuous [Mean (Standard Deviation); unit: years] — All subjects who underwent an implant attempt (186) were included in the study population analyses.
  years | 69.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects who underwent an implant attempt (186) were included in the study population analyses.
  Participants
    Female | 48
    Male | 138
Region of Enrollment [Number; unit: participants]
  United States | 143
  Canada | 43
New York Heart Association [Number; unit: Participants] — All subjects who underwent an implant attempt (186) were included in the study population analyses. Some subjects did not report data or data was outside the criteria, this was captured as a protocol deviation.
  Participants
    Class III | 182
    Class IV | 2
    Missing | 2
Race / Ethnicity [Number; unit: Participants] — All subjects who underwent an implant attempt (186) were included in the study population analyses.
  Participants
    American Indian or Alaska Native | 1
    Asian | 2
    Black or African American | 10
    Columbian | 1
    Hispanic or Latino | 3
    Native Hawaiian or Pacific Islander | 1
    Sri Lankan | 1
    Subject chose not to provide | 6
    White | 161
Intrinsic QRS Width [Mean (Standard Deviation); unit: Milliseconds] — All subjects who underwent an implant attempt (186) were included in the study population analyses. Some subjects did not report data or data was outside the criteria, this was captured as a protocol deviation.
  Milliseconds | 153.1 (24.1)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percent] — All subjects who underwent an implant attempt (186) were included in the study population analyses. Some subjects did not report data or data was outside the criteria, this was captured as a protocol deviation. Left ventricular ejection fraction is the fraction of blood pumped out of the left ventricle with each heartbeat. For this measurement, the fraction is presented as a percent.
  Percent | 24.2 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Safety (Subjects Without a Model 4196 Lead Related Complication)
Description: A subject who was free of a Model 4196 lead related complication by one month visit.
Time Frame: One Month
Population: Subjects who underwent a Model 4196 left ventricular (LV) lead implant attempt and completed 1-month visit; or experienced Model 4196 lead related complications by 1-month visit.
Measure: Number; unit: participants
Groups:
- 4196 Lead: Subjects who underwent Model 4196 left ventricular lead implant attempt
Arm/Group | 4196 Lead
Number analyzed (Participants) | 176
participants | 168 [92 to 100]
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample proportion = 0.955, 95% CI [0.92 to 0.955] — 1-side 95% confidence limit lower bound

2. Secondary Outcome: Subjects Successfully Implanted With Model 4196 Lead
Description: A successful implant occurs when the Model 4196 lead is implanted in the left ventricle of the heart and functions appropriately.
Time Frame: Implant
Population: Subjects who underwent Model 4196 lead implant attempt.
Measure: Number; unit: participants
Groups:
- 4196 Lead: Subjects who underwent Model 4196 LV lead implant attempt
Arm/Group | 4196 Lead
Number analyzed (Participants) | 177
participants | 170
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample proportion = 0.96, 95% CI [0.932 to 0.989]

3. Primary Outcome: Efficacy (Pacing Voltage Thresholds of Distal Tip Electrode)
Description: Model 4196 lead distal tip electrode mean pacing voltage threshold (at 0.5 milliseconds [ms])
Time Frame: One Month
Population: Subjects with pacing threshold at tip electrode captured at 0.5 milliseconds (ms) at 1-month visit.
Measure: Mean (Standard Deviation); unit: volts
Groups:
- 4196 Lead: Subjects with tip electrode threshold capture at 0.5ms at 1-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 160
volts | 1.1 (0.9)
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample mean = 1.1, 95% CI [1.1 to 1.2], Standard Deviation 0.9 — 1-side 95% confidence limit upper bound

4. Primary Outcome: Efficacy (Pacing Voltage Threshold of Proximal Ring Electrode)
Description: Model 4196 lead proximal ring electrode mean pacing voltage threshold (at 0.5 milliseconds [ms])
Time Frame: Three Months
Population: Subjects with pacing threshold at ring electrode captured at 0.5 milliseconds (ms) at 3-month visit.
Measure: Mean (Standard Deviation); unit: volts
Groups:
- 4196 Lead: Subjects with ring electrode threshold captured at 0.5ms at 3-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 135
volts | 1.9 (2.0)
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample mean = 1.9, 97.5% CI [1.9 to 2.2], Standard Deviation 2.0 — 1-sided 97.5% confidence limit upper bound

5. Secondary Outcome: Subjects Successfully Implanted After Cannulation
Description: A successful implant occurs when the coronary sinus (CS) is successfully cannulated and a left ventricular lead is implanted in the left ventricle of the heart and functions appropriately.
Time Frame: Implant
Population: Subjects with successful CS cannulation after an incision was made (implant attempt)
Measure: Number; unit: participants
Groups:
- 4196 Lead: Subjects who underwent an implant attempt with successful CS cannulation
Arm/Group | 4196 Lead
Number analyzed (Participants) | 183
participants | 181
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample proportion = 0.989, 95% CI [0.974 to 1]

6. Secondary Outcome: All Left Ventricular Leads
Description: All left ventricular leads successfully implanted
Time Frame: Implant
Population: Subjects who underwent an implant attempt.
Measure: Number; unit: participants
Groups:
- 4196 Lead: Subjects who underwent an implant attempt
Arm/Group | 4196 Lead
Number analyzed (Participants) | 186
participants | 181
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample proportion = 0.973, 95% CI [0.950 to 0.996]

7. Secondary Outcome: All Medtronic Left Ventricular Leads (Attain Family)
Description: All Medtronic left ventricular leads (Lead Model Numbers included 4193, 4194, 4195 and 4196) successfully implanted
Time Frame: Implant
Population: Subjects who underwent an implant attempt.
Measure: Number; unit: participants
Arm/Group | 4196 Lead
Number analyzed (Participants) | 186
participants | 181
Statistical Analysis 1: Comparison: 4196 Lead; Test type: Superiority or Other; One sample proportion = 0.973, 95% CI [0.950 to 0.996]

8. Secondary Outcome: Cannulation Time
Description: Cannulation time was defined as the time from insertion of the first CS cannulation catheter to the first CS cannulation.
Time Frame: Implant
Population: Subjects successfully implanted with a Model 4196 lead.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 4196 Lead: Subjects successfully implanted with a Model 4196 lead
Arm/Group | 4196 Lead
Number analyzed (Participants) | 170
minutes | 10.4 (4.0)

9. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time was defined as the total time the fluoroscope was imaging.
Time Frame: Implant
Population: Subjects successfully implanted with a Model 4196 lead.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 4196 Lead
Number analyzed (Participants) | 170
minutes | 25.2 (18.9)

10. Secondary Outcome: Model 4196 Lead Placement Time
Description: Model 4196 lead placement time was defined as the time from insertion of the successfully placed lead to the time when it was placed in the first acceptable pacing location.
Time Frame: Implant
Population: Subjects successfully implanted with a Model 4196 lead.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 4196 Lead
Number analyzed (Participants) | 170
minutes | 11.9 (10.0)

11. Secondary Outcome: Total Implant Time
Description: Total implant time was defined as time from initial incision to final closure.
Time Frame: Implant
Population: Subjects successfully implanted with a Model 4196 lead.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 4196 Lead
Number analyzed (Participants) | 170
minutes | 117.1 (101.5)

12. Secondary Outcome: Assessment of Lead Handling Characteristics
Description: Lead handling characteristics assessed as "acceptable" by physicians
Time Frame: Implant
Population: All available assessments from physicians.
Measure: Number; unit: participants
Arm/Group | 4196 Lead
Number analyzed (Participants) | 177
participants | 174

13. Secondary Outcome: Electrical Performance - Tip Electrode: Sensing
Description: Model 4196 lead tip electrode R-wave amplitude
Time Frame: 12-month
Population: Subjects with Model 4196 lead implanted and an intrinsic R-wave available at 12-month visit.
Measure: Mean (Standard Deviation); unit: millivolt (mV)
Groups:
- 4196 Lead: Subjects with tip electrode R-wave amplitude at 12-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 121
millivolt (mV) | 17.0 (5.9)

14. Secondary Outcome: Electrical Performance - Tip Electrode: LV Voltage Threshold
Description: Model 4196 lead tip electrode LV voltage threshold
Time Frame: 12-month
Population: Subjects with Model 4196 lead implanted and 12-month visit completed.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- 4196 Lead: Subjects with tip electrode threshold captured at 0.5ms at 12-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 131
Volts | 1.2 (1.0)

15. Secondary Outcome: Electrical Performance -Tip Electrode: Pacing Impedance
Description: Model 4196 lead tip electrode pacing impedance
Time Frame: 12-month
Population: Subjects with Model 4196 lead implanted and 12-month visit completed.
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- 4196 Lead: Subjects with tip electrode pacing impedance at 12-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 133
Ohms | 508.7 (144.5)

16. Secondary Outcome: Electrical Performance -Ring Electrode: Sensing
Description: Model 4196 lead ring electrode R-wave amplitude
Time Frame: Implant
Population: Subjects with Model 4196 lead implanted and with intrinsic R-wave amplitude at implant.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- 4196 Lead: Subjects with ring electrode R-wave amplitude at implant
Arm/Group | 4196 Lead
Number analyzed (Participants) | 162
mV | 15.4 (6.9)

17. Secondary Outcome: Electrical Performance - Ring Electrode: LV Voltage Threshold
Description: Model 4196 lead ring electrode LV voltage threshold
Time Frame: 12-month
Population: Subjects with Model 4196 lead implanted and 12-month visit completed.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- 4196 Lead: Subjects with ring electrode threshold captured at 0.5ms at 12-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 115
Volts | 2.0 (2.0)

18. Secondary Outcome: Electrical Performance -Ring Electrode: Pacing Impedance
Description: Model 4196 lead ring electrode pacing impedance
Time Frame: 12-Month
Population: Subjects with Model 4196 lead implanted and completed 12-month visit.
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- 4196 Lead: Subjects with ring electrode pacing impedance at 12-month
Arm/Group | 4196 Lead
Number analyzed (Participants) | 133
Ohms | 497.1 (262.9)

19. Secondary Outcome: Summarize All Adverse Events
Description: All adverse events were collected for this trial such as, but not limited to, the following: Atrial Fibrillation, Chest Pain, Pneumonia, Cold/Flu
Time Frame: Up to 18 months
Population: All subjects enrolled into the 4196 study.
Measure: Number; unit: adverse events
Groups:
- 4196 Lead: All enrolled subjects
Arm/Group | 4196 Lead
Number analyzed (Participants) | 190
adverse events | 538

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Medtronic reviews publications to determine if confidential information ("CI") is included. Any such CI is deleted before publication. Medtronic may not censor/interfere with the publication. Investigators may publish single-site publications after a decision by Medtronic that no multi-site study publication will be done or 12 months after the study is closed, whichever is earlier.